CLINICAL TRIAL: NCT01639105
Title: 10 600 nm Ablative Fractional Laser Treatment of Scars: a Prospective Single Blinded Within Patient Controlled Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/395
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Scars After Surgical Intervention
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- treated half of the scar (Experimental)
  Interventions: Procedure: Laser treatment
- untreated half of the scar (No Intervention)

INTERVENTIONS:
Procedure: Laser treatment — 10 600 NM ABLATIEVE FRACTIONATED LASER
  Arms: treated half of the scar

SUMMARY:
Rationale The cosmetic aspect of scars is a frequent reason for consultation. It plays an important role in patient satisfaction and self-image. Several treatment modalities are proposed for scars with variable success.

Ablative fractional laser treatment is a rather new concept. Many microscopic small laser beams target the dermis in a grid pattern. The vertical columns of skin hit by the laser beams heat up. This thermal effect stimulates the wound healing and potentially leads to a remodeling of the skin structure.

Ablative fractional laser treatment has been used successfully for treatment of pigment changes, wrinkles, acne scars and thermal burn wounds. It has been reported that CO2 ablative fractional laser treatment has a positive clinical effect on various types of scars however this has not been proven yet in a prospective randomized trial. The low morbidity of the treatment and the lack of convincing adapted treatment modalities for various types of scars make this treatment attractive.

That's why the investigators aim with this randomized study to evaluate the clinical effect and the safety of 10 600 nm ablative fractional laser therapy for patients with recent scars due to surgical interventions.

Goal Evaluate the efficacy of three 10 600 nm ablative fractional laser treatments for the above mentioned scars, three months after the last laser treatment, with a prospective randomized intra-patient controlled study.

Study design Prospective single blinded randomized intra-patient controlled study. The study comprises 4 study visits.

Study population The population consists of one group of patients with scars after recent surgical operations. The patients must meet the inclusion and exclusion criteria described in the protocol.

Method The scar will be divided in two equal halves. The two halves will be randomized. One part will not be treated. The other part will undergo three times the 10 600 nm ablative laser therapy with 4 weeks interval between the treatments. The efficacy of the treatment will be evaluated three months after the last treatment with objective and subjective parameters.

Most important study endpoints:

* Evaluation of the efficacy of the treatment. A blinded clinical scar evaluation will be done of the treated and untreated parts with the POSAS scar scale, by a study collaborator and by the patient himself, on a category scale of 0 to 10 (0 = normal skin, 10 = worst scar imaginable), before start and twelve weeks after the last treatment.
* Evaluation of the pain related to the treatment. The pain will be scored by the patient with the VAS category scale from 0 to 10 (0 = no pain, 10 = worst pain ever).
* Evaluation of the side effects of the treatment. A standardized form will be used.
* Evaluation of the global patient satisfaction regarding the treatment.
* Clinical photos, before start and twelve weeks after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Scars caused by surgical intervention, that are 2 months old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical aspect of the scar 3 months after the last laser treatment | 3 months after the last laser treatment
  POSAS scar scale

SECONDARY OUTCOMES:
Pain | 3 months after the last laser treatment
  VAS scale for pain measurement
Number and severity of side effects | 3 months after the last laser treatment
  Will be measured by clinical photographs
satisfaction | 3 months after the last laser treatment
  Will be measured with the standardized satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Boone, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium